CLINICAL TRIAL: NCT03098030
Title: A Two-part, Open-label, Randomized, Phase 2/3 Study of Dinutuximab and Irinotecan Versus Irinotecan for Second Line Treatment of Subjects With Relapsed or Refractory Small Cell Lung Cancer
Brief Title: Dinutuximab and Irinotecan Versus Irinotecan to Treat Subjects With Relapsed or Refractory Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIV-SCLC-301
Record Dates: First submitted 2017-03-22; First posted 2017-03-31 (Actual); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Small Cell Lung Cancer
Keywords: Dinutuximab; Irinotecan; Topotecan
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — dinutuximab; Irinotecan; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Dinutuximab + Irinotecan (Experimental): Dinutuximab (10 mg/m^2 IV) + Irinotecan (350 mg/m^2 IV) on Day 1 of every 21 days (q21d). Dinutuximab dose will be escalated in 2 mg/m^2 increments per cycle if maximal pain is <Grade 2 (and without opioids) and otherwise tolerated, up to a maximum dose of 17.5 mg/m^2 IV.
  Interventions: Biological: Dinutuximab; Drug: Irinotecan
- Part 2: Irinotecan (Active Comparator): Irinotecan (350 mg/m^2 IV) on Day 1 of each q21d cycle.
  Interventions: Drug: Irinotecan
- Part 2: Dinutuximab + Irinotecan (Experimental): Dinutuximab (16 mg/m^2 IV) + Irinotecan (350 mg/m^2 IV) on Day 1 of each q21d cycle. Dinutuximab dose will be escalated in 2 mg/m^2 increments per cycle if maximal pain is <Grade 2 (and without opioids) and otherwise tolerated, up to a maximum dose of 17.5 mg/m^2 IV.
  Interventions: Biological: Dinutuximab; Drug: Irinotecan
- Part 2: Topotecan (Active Comparator): Topotecan (1.5 mg/m^2 IV) on Days 1 to 5 of each q21d cycle.
  Interventions: Drug: Topotecan

INTERVENTIONS:
Biological: Dinutuximab — Dinutuximab injection, for intravenous (IV) use
  Other Names: Unituxin®; ch14.18
  Arms: Part 1: Dinutuximab + Irinotecan; Part 2: Dinutuximab + Irinotecan
Drug: Irinotecan — Irinotecan injection, IV infusion
  Other Names: Camptosar®
  Arms: Part 1: Dinutuximab + Irinotecan; Part 2: Dinutuximab + Irinotecan; Part 2: Irinotecan
Drug: Topotecan — Topotecan for injection
  Other Names: Hycamtin®
  Arms: Part 2: Topotecan

SUMMARY:
This is a 2-part, multicenter, open-label, randomized study of dinutuximab and irinotecan versus irinotecan alone in subjects with relapsed or refractory small cell lung cancer (SCLC). Part 1 of the study involves intrasubject dose escalation to evaluate the safety and tolerability of dinutuximab in combination with irinotecan. Part 2 of the study is designed to determine whether dinutuximab plus irinotecan prolongs overall survival (OS) compared with irinotecan alone. Subjects in Part 2 will be randomized in a 2:2:1 fashion to 1 of 3 treatment groups: (A) irinotecan; (B) dinutuximab plus irinotecan; or (C) topotecan. Randomization will be stratified by duration of response to prior platinum therapy (relapse-free period <3 months or ≥3 months).

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically confirmed SCLC (undifferentiated small-cell carcinoma arising in or consistent with lung cancer origin).
2. Documented relapse or disease progression during or after first-line platinum-based therapy (subjects refractory to initial platinum-based therapy are eligible).
3. Have no curative therapy available.
4. Have a life expectancy of at least 12 weeks.
5. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Have adequate bone marrow and hepatic function.
7. Have calculated creatinine clearance (CrCL) ≥30 mL/minute or serum creatinine ≤1.5 times below the upper limit of normal.
8. Women of reproductive potential must not be pregnant or breastfeeding and have a negative urine or serum pregnancy test obtained within 7 days prior to the first dose of study treatment.
9. Subjects must agree to consistently use 2 forms of highly effective contraception/birth control between signing of the informed consent and 60 days after the last study drug administration.

Exclusion Criteria:

1. Candidate for re-treatment with original platinum-based regimen as second-line therapy.
2. Prior treatment with irinotecan, topotecan, or dinutuximab.
3. Have active brain metastases. Subjects with brain metastases are allowed if they completed definitive brain therapy, are asymptomatic and radiologically stable, and if they are not currently receiving corticosteroids or radiation.
4. Have mixed small cell and non-small cell histologic features.
5. Have a previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study, except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta and Tis [carcinoma in situ]) or any previous cancer curatively treated <3 years ago.
6. Have a history or current evidence of uncontrolled cardiovascular disease.
7. Have not recovered from prior surgery, significant trauma, systemic anticancer therapy, radiation therapy or investigational therapy to Grade 1 or better toxicity prior to enrollment (Part 1) or randomization (Part 2).
8. Have had organ allograft or hematopoietic transplantation.
9. Known to be human immunodeficiency virus (HIV) positive.
10. Have an active infection requiring treatment or one that is clinically serious in the Investigator's opinion.
11. Have received a live vaccine within 6 months of enrollment (Part 1) or randomization (Part 2).
12. Exposure to strong CYP3A4 and/or UGT1A1 inhibitors and strong CYP3A4 inducers within 14 days of enrollment (Part 1) or randomization (Part 2).
13. Have any clinical condition that is considered unstable or might jeopardize the safety of the subject and/or influence the subject's compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (225):
- United States (40):
  - Alaska Clinical Research Center, Anchorage, Alaska
  - Cancer Treatment Centers of America - Western Regional Medical Center, Goodyear, Arizona
  - Innovative Clinical Research Institute, Tucson, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Olive View - UCLA, Sylmar, California
  - Innovative Clinical Research Institute, Whittier, California
  - Hartford Hospital, Hartford, Connecticut
  - Eastern Connecticut Hematology and Oncology Assoc, Norwich, Connecticut
  - Alpha Oncology Research LLC, DeBary, Florida
  - 21st Century Oncology, Jacksonville, Florida
  - Comprehensive Hematology Oncology, St. Petersburg, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - Baptist Health Floyd Cancer Center, New Albany, Indiana
  - Physicians' Clinic of Iowa Hematology and Oncology, Cedar Rapids, Iowa
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - 21st Century Oncology, Louisville, Kentucky
  - Cox Health Medical, Springfield, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - The University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - UH Cleveland Medical Center, Cleveland, Ohio
  - Cancer Treatment Centers of America at Southwestern RMC, Tulsa, Oklahoma
  - Kaiser Permanente Northwest Center for Health Research CRSS, Portland, Oregon
  - Fox Chase Cancer Center Office of Clinical Research, Philadelphia, Pennsylvania
  - Cancer Treatment Centers of America at Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Charleston Oncology, Charleston, South Carolina
  - Spartanburg Medical Center/Gibbs Cancer Center and Research Institute, Spartanburg, South Carolina
  - Prairie Lakes Health Care, Watertown, South Dakota
  - Center for Biomedical Research, Knoxville, Tennessee
  - Texas Health Physicians Group, Arlington, Texas
  - Plano Cancer Institute, Plano, Texas
  - The University of Texas Health Science Center at Tyler, Office of Clinical Studies, Tyler, Texas
  - Vista Oncology (Shelton office), Shelton, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - Camden Clark Medical Center / Regional Cancer Center, Parkersburg, West Virginia
  - University of Wisoncsin - Carbone Cancer Ctr, Madison, Wisconsin
- Australia (4):
  - Mid North Coast Cancer Institute Coff Habour Health Campus, Coffs Harbour, New South Wales
  - Mater Misericordiae Limited and Mater Medical Research Institute Limited, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Ballarat Health Services, Ballarat, Victoria
- Bulgaria (14):
  - Medical Oncology Department, Specialized Hospital for Active Treatment of Oncology Sveti Mina EOOD - Blagoevgrad, Blagoevgrad
  - Department of Medical Oncology, Complex Oncology Center - Burgas EOOD, Burgas, Burgas
  - Medical Oncology Department, Multiprofile Hospital for Active Treatment - Dobrich AD, Dobrich, Dobrich
  - Medical Oncology Department, Multiprofile Hospital for Active Treatment - Dr. Tota Venkova AD, Gabrovo, Gabrovo
  - Medical Oncology Department, Multiprofile Hospital for Active Treatment - Uni Hospital OOD, Panagiurishte, Panagyurishte
  - Clinic of Oncology, UMHAT Dr. Georgi Stranski - Pleven, Pleven
  - Clinic of Oncology, UMHAT Pulmed, Plovdiv
  - First Department of Medical Oncology, Gastroenterology and Pulmology, Complex Oncology Center - Plovdiv EOOD, Plovdiv
  - First Department for Medical Oncology, Multiprofile Hospital for Active Treatement Serdika EOOD, Sofia, Sofia
  - Medical Oncology Clinic, Multiprofile Hospital for Active Treatment (MHAT) for Female's Health - Nadezhda OOD, Sofia, Sofia
  - Medical Oncology Department, University Multiprofile Hospital for Active Treatment Sv. Ivan Rilski EAD, Sofia, Sofia
  - Clinic for Chemotherapy, Specialized Hospital for Active Treatment in Oncology EAD, Sofia, Sofia
  - Clinic of Oncology, UMHAT SofiaMed, Sofia
  - Clinic of Oncology, MHAT Sveta Marina, Varna
- Canada (6):
  - Cross Cancer Institute - Clinical Trials Unit, Edmonton, Alberta
  - Horizon Health Network - The Moncton Hosoital, Moncton, New Brunswick
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Windsor Regional Hospital Cancer Program, Windsor, Ontario
  - McGill University Health Center, Montreal, Quebec
  - L'Institut Universitaire de Cardiologie et de pneumologie de Quebec, Québec, Quebec
- France (14):
  - Hopital Nord, Marseille, Alpes-Côte d'Azur
  - URCOT : Unité de Recherche Commune en Oncologie Thoracique Service de pneumologie de l'hôpital de la Croix-Rousse, Bron, Auvergne-Rhône-Alpes
  - URCOT : Unité de Recherche Commune en Oncologie Thoracique Service de pneumologie de l'hôpital de la Croix-Rousse, Lyon, Auvergne-Rhône-Alpes
  - Service de Pneumologie aiguë et Cancérologie Thoracique Centre hospitalier Lyon-Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Institut Regional du Cancer de Montpellier, Montpellier, Occitanie
  - Institut de Cancérologie de l'Ouest - Centre Paul Papin, Angers, Pays de la Loire Region
  - Clinique Victor Hugo, Le Mans, Pays de la Loire Region
  - CHU Brest, Brest
  - Centre François Baclesse, Caen
  - CHI Créteil, Créteil
  - Institut Paoli-Calmettes, Service Dòncologie Médicale, Marseille
  - Institut de Cancérologie de l'Ouest - Centre René Gauducheau, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Nouvel Hôpital Civil de Strasbourg, Strasbourg
- Georgia (5):
  - LTD High Technology Hospital Medcenter, Batumi
  - LTD ''Accad. F. Todua Medical Center-Research Institute of Clinical Medicine'', Tbilisi
  - High Technology Medical Center, University Clinic, Tbilisi
  - Institute of Clinical Oncology, Tbilisi
  - Multiprofile Clinic Consillium Medulla, Tbilisi
- Hong Kong (3):
  - Princess Margaret Hospital, Kowloon
  - Queen Elizabeth Hospital, Kowloon
  - Queen Mary Hospital, Pokfulam
- Hungary (11):
  - Hetenyi Geza Hospital, Szolnok, Jász-Nagykun-Szolnok
  - Koranyi National Institute of Pulmonology - Horváth, Budapest
  - Koranyi National Institute of TBC and Pulmonology, Budapest
  - Korányi National Institute, Budapest
  - Semmelweis Egyetem AOK Pulmonologiai Klinika, Budapest
  - Veszprém Megyei Tüdőgyógyintézet, Farkasgyepű
  - Matrai Gyogyintezet, Mátraháza
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktatókórház, Semmelweis Tagkórház, Tüdőgyógyászati Osztály, Miskolc
  - Komarom-Esztergom Megyei Onkorm. Szent Borbala Korhaza, Tatabánya
  - Tudogyogyintezet Torokbalint, Törökbálint
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg
- India (8):
  - Sri Venkateshwara Hospitals, Bangalore, Karnataka
  - KLES Dr Prabhakar Kore Hospital & MRC, Nehru Nagar, Karnataka
  - Jaslok Hospital & Research Center, Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital, Pune, Maharashtra
  - Grant Medical Foundation Ruby Hall Clinic, Pune, Maharashtra
  - Birla Cancer Centre, SMS Hospital, Jaipur, Rajasthan
  - Healthcare Global (HCG) Towers, Bangalore
  - Bhagawan Mahaveer Cancer Hospital, Jaipur
- Italy (7):
  - Dipartimento di Oncologia, ARNAS Garibaldi, Catania
  - Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia (IEO), Milano, Milan
  - Ospedale Santa Maria della Misericordia, Perugia, Perugia
  - Radiation Oncology, Campus Bio-Medico University, Rome
  - Division of Medical Oncology and Immunotherapy, Department of Oncology, University Hospital of Siena, Siena
  - A.O.U. San Luigi Gonzaga, Orbassano (Torino), Torino
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences (LSMU) Kauno Klinikos, Kaunas
  - National Cancer Institute, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Malaysia (4):
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Department of Medicine, Faculty of Medicine, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching
  - National Cancer Institute, Putrajaya
- Philippines (5):
  - Cebu Doctors University Hospital, Cebu City
  - Davao Doctors Hospital, Davao City
  - Manila Doctors Hospital, Manila
  - St. Luke's Medical Center - Quezon City, Quezon City
  - St. Luke's Medical Centre, Quezon City
- Poland (9):
  - Szpital Specjalistyczny w Prabutach Sp. z o.o, Prabuty, Pomeranian Voivodeship
  - Samodzielny Publiczny Zespół Gruźlicy i Chorób Płuc w Olsztynie, Olsztyn, Warmian-Masurian Voivodeship
  - Samodzielny Specjalistyczny ZespółZakładów Opieki Zdrowotnej im. dr. Teodora Dunina, Mrozy
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock
  - Szpital Chorób Płuc im Św. Józefa w Pilchowicach, Pilchowice
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii im. Eugenii i Janusza Zeylandów, Poznan
  - Centrum Onkologii-Instytut im. Sklodowskiej-Curie, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska sp. komandytowo-akcyjna, Lodz, Łódź Voivodeship
- Romania (8):
  - Oncopremium Team LTD, Baia Mare
  - Institute of Oncology Prof. Dr. I.Chiricuta Cluj-Napoca, Cluj-Napoca
  - Medisprof LTD, Cluj-Napoca
  - SC Oncolab LTD, Craiova
  - SC Oncology Center Sf. Nectarie LTD, Craiova
  - Emergency County Hospital Satu-Mare, Medical Oncology Clinic, Satu Mare
  - Emergency Hospital ,Sf. Ioan cel Nou', Suceava
  - Oncocenter Oncology Clinic LTD, Timișoara
- Russia (18):
  - State Budgetary Healthcare Institution of Arkhangelsk Region Arkhangelsk Clinical Oncology Dispensary, Arkhangelsk
  - Region Budgetary Healthcare Institution, Kursk Regional Clinical Oncology Dispensary of Healthcare Committee of Kursk Region, Kursk
  - Federal State Budgetary Institution, Natiоnal Medical Research Center of Oncology n.a. N.N. Blokhin of Ministry of Healthcare of the Russian Federation, Moscow
  - State Budgetary Healthcare Institution of Moscow, Moscow City Oncology Hospital #62 of Moscow Healthcare Department, Moscow
  - State Budgetary Healthcare Institution of Arkhangelsk region "Arkhangelsk Clinical Oncology Dispensary", Moscow
  - State Budgetary Healthcare Institution of Novosibirsk Region, Сity Clinical Hospital #1, Novosibirsk
  - State Budgetary Healthcare Institution of Novosibirsk Region, Novosibirsk Regional Oncology Dispensary, Novosibirsk
  - Budgetary Healthcare Institution of Omsk Region, Clinical Oncology Dispensary, Omsk
  - State Budgetary Healthcare Institution, Orenburg Regional Clinical Oncology Dispensary, Orenburg
  - State Budgetary Healthcare Institution, Leningrad Regional Clinical Hospital, Saint Petersburg
  - Center of Palliative Care-Devita LLC, Saint Petersburg
  - BioEq, LLC, Saint Petersburg
  - Federal State Budgetary Institution, Scientific Research Institute of Oncology n.a. Petrov, Saint Petersburg
  - State Budgetary Healthcare Institution, Saint-Petersburg Clinical Scientific Practical Center of Specialized Kinds of Medical Care (Oncological), Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution, City Clinical Oncology Dispensary, Saint Petersburg
  - State Budgetary Healthcare Institution, Samara Regional Clinical Oncology Dispensary, Samara
  - State Budgetary Healthcare Institution of Yaroslavl Region, Regional Oncology Hospital, Yaroslavl
  - State Budgetary Healthcare Institution of Sverdlovsk Region, Sverdlovsk Regional Oncology Dispensary, Yekaterinburg
- Slovakia (2):
  - St. Jacob´s Hospital Bardejov - Department of Clinical Oncology, Bardejov
  - Faculty Hospital Zilina, Žilina
- South Korea (16):
  - Kosin University Gospel Hospital, Busan
  - Chungbuk National University Hospital, Chungcheongbuk-do
  - Kyungpook National University Medical Center, Daegu
  - Kyungpook University Chilgok Hospital, Daegu
  - Keimyung University Dongsan Medical Centre, Daegu
  - Chungnam National University Hospital, Daejeon
  - CHA Bundang Medical Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Inha University Hospital, Incheon
  - Chonnam National University Hwasun Hospital, Jeonnam
  - Gachon Universtiy Gil Medical Center, Namdong
  - Korea University Anam Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wonju-Si, Gangwon-do
- Spain (23):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - CHU A Coruña, A Coruña, Galicia
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital General de Alicante, Alicante
  - Hospital Quirón Dexeus, Barcelona
  - Hospital Universitari Vall d´Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Instituto Catalán de Oncología (ICO) - Josep Trueta, Girona
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital General Universitário Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Madrid Norte Sanchinarro, Madrid
  - H. M. Puerta del Sur (H. Móstoles), Madrid
  - Hospital Regional de Málaga (H. Carlos Haya), Málaga
  - Complexo Hospitalario Universitario de Ourense (CHUO), Ourense
  - Hospital Virgen de los Lirios Alcoy, Planta
  - Corporació Sanitària Parc Taulí, Sabadell
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario y Politécnico de La Fe, Valencia
  - Hospital Álvaro Cunqueiro, Vigo
  - Hospital Lozano Blesa, Zaragoza
- Taiwan (5):
  - E-Da Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Chi Mei Hospital, Liouying, Tainan
  - Chang-Gung Memorial Hospital, Linkou, Taoyuan
- Thailand (7):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - National Cancer Institute of Thailand, Bangkok
  - Siriraj Hopsital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Naresuan University Hospital, Phitsanulok
  - Songklanagarind Hospital, Songkhla
- Ukraine (6):
  - Municipal Non-profit Enterprise "City Clinical Hospital #4" of Dnipro City Council," Municipal Institution "Multifield Dnipropetrovsk City Hospital #4" of Dnipropetrovsk Regional Council, Department of Chemotherapy, Dnipro, Dnipropetrovsk Oblast
  - Municipal Nonprofit Institution "Cental Municipal Clinical Hospital" of Uzhgorod City Council, Municipal Oncology Centre, Uzhhorod, Zakarpattia Oblast
  - Regional Communal Nonprofit Enterprise, Municipal Institution Chernivtsi Regional Clinical Oncology Dispensary, Surgery Department, State Higher Educational Establishment of Ukraine, Bukovinian State Medical University, Department of Onc and Radiology, Chernivtsi
  - Communal Non-profit Enterprise "Kyiv City Clinical Oncology Center" of Executive body of Kyiv City Council, Kyiv City Clinical Oncology Center by Main Department of Health Protection Kyiv, Hospital of Day Stay for Oncology Patients, Kiev
  - Municipal Nonprofit Institution "Odessa Regional Oncology Dispensary" of Odessa Regional Council, Municipal Institution Odesa Regional Oncology Dispensary, Hospital of Day Stay (Unit of Dispensary-Polyclinic Department), Odesa
  - Municipal Nonprofit Institution "Podilsky Regional Oncology Center" of Vinnytsa City Council, Podilsky Regional Oncology Сenter, Department of Chemotherapy, Vinnitsya
- United Kingdom (7):
  - Princess Alexandra Hospital, Harlow, Essex
  - Royal Marsden Hospital, Chelsea, London
  - St James' Institute of Oncology, Leeds
  - St Bartholomew's Hospital, London
  - Royal Free Hospital, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edelman MJ, Dvorkin M, Laktionov K, Navarro A, Juan-Vidal O, Kozlov V, Golden G, Jordan O, Deng CQ, Bentsion D, Chouaid C, Dechev H, Dowlati A, Fernandez Nunez N, Ivashchuk O, Kiladze I, Kortua T, Leighl N, Luft A, Makharadze T, Min Y, Quantin X; DISTINCT study investigators. Randomized phase 3 study of the anti-disialoganglioside antibody dinutuximab and irinotecan vs irinotecan or topotecan for second-line treatment of small cell lung cancer. Lung Cancer. 2022 Apr;166:135-142. doi: 10.1016/j.lungcan.2022.03.003. Epub 2022 Mar 4. PMID 35278766

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Dinutuximab + Irinotecan: Dinutuximab (10 mg/m^2 IV) + Irinotecan (350 mg/m^2 IV) on Day 1 of every 21 days (q21d). Dinutuximab dose will be escalated in 2 mg/m^2 increments per cycle if maximal pain is <Grade 2 or Grade 2/3 that in the view of the Investigator is adequately managed and otherwise tolerated, up to a maximum dose of 17.5 mg/m^2 IV.
  Dinutuximab: Dinutuximab injection, for intravenous (IV) use
  Irinotecan: Irinotecan injection, IV infusion
- Part 2: Dinutuximab + Irinotecan: Dinutuximab (16 mg/m^2 IV) + Irinotecan (350 mg/m^2 IV) on Day 1 of each q21d cycle. Dinutuximab dose will be escalated in 2 mg/m^2 increments per cycle if maximal pain is <Grade 2 or Grade 2/3 that in the view of the Investigator is adequately managed and otherwise tolerated, up to a maximum dose of 17.5 mg/m^2 IV.
  Dinutuximab: Dinutuximab injection, for intravenous (IV) use
  Irinotecan: Irinotecan injection, IV infusion
Period: Overall Study
Arm/Group | Part 1: Dinutuximab + Irinotecan | Part 2: Dinutuximab + Irinotecan | Part 2: Irinotecan | Part 2: Topotecan
Started | 12 | 187 | 190 | 94
Completed | 2 (Represents number of subjects that had not discontinued the study at time of data lock.) | 24 (Represents number of subjects that had not discontinued the study at time of data lock.) | 24 (Represents number of subjects that had not discontinued the study at time of data lock.) | 9 (Represents number of subjects that had not discontinued the study at time of data lock.)
Not Completed | 10 | 163 | 166 | 85
Not completed — Death | 10 | 156 | 156 | 82
Not completed — Withdrawal by Subject | 0 | 7 | 8 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Dinutuximab + Irinotecan | Part 2: Dinutuximab + Irinotecan | Part 2: Irinotecan | Part 2: Topotecan | Total
Number analyzed (Participants) | 12 | 187 | 190 | 94 | 483
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (8.8) | 61.3 (8.7) | 61.5 (9.0) | 62.5 (8.4) | 61.6 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 45 | 43 | 26 | 118
  Male | 8 | 142 | 147 | 68 | 365
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 2 | 4 | 11
  Not Hispanic or Latino | 4 | 137 | 142 | 72 | 355
  Unknown or Not Reported | 8 | 45 | 46 | 18 | 117
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 28 | 34 | 18 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3 | 6
  White | 4 | 113 | 106 | 54 | 277
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 8 | 45 | 47 | 19 | 119
Region of Enrollment [Count of Participants; unit: Participants]
  Southeast Asia | 0 | 27 | 39 | 16 | 82
  North America | 4 | 31 | 32 | 16 | 83
  Europe | 8 | 129 | 119 | 62 | 318
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Performance Status was used as a measure of how the disease impacted the patient's daily living abilities with eligible grading levels defined as follows:
  0 = Fully active, able to carry on all pre-disease performance without restriction
  1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    Performance Status = 0 | 3 | 37 | 40 | 19 | 99
    Performance Status = 1 | 9 | 150 | 150 | 75 | 384
Tobacco Use [Count of Participants; unit: Participants]
  No | 0 | 22 | 12 | 12 | 46
  Yes | 12 | 165 | 178 | 82 | 437
Body Surface Area (m^2) [Mean (Standard Deviation); unit: m^2] | 26.40 (4.42) | 25.84 (5.01) | 25.95 (4.91) | 25.54 (4.89) | 25.82 (4.94)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS will be derived as: (date of death - date of randomization) + 1. Subjects who are alive or permanently lost to follow-up at the cut-off date for the analysis will be censored at the last date the subject was known to be alive.
Time Frame: Up to approximately 2.5 years
Population: The analysis population was based on the Intent to Treat (ITT) Analysis Set, which per the Statistical Analysis Plan was defined as all subjects randomized in Part 2 of the study, as assigned to treatment (i.e., n = 471). As such, these results do not include the subjects enrolled in Part 1 of the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Dinutuximab + Irinotecan | Part 2: Irinotecan | Part 2: Topotecan
Number analyzed (Participants) | 187 | 190 | 94
months | 6.9 [6.0 to 7.6] | 7.0 [5.6 to 8.9] | 7.4 [6.1 to 9.3]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS will be defined as the time from the date of randomization to the date of first documentation of tumor progression or death from any cause, whichever occurs first.
Time Frame: Up to approximately 2.5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Dinutuximab + Irinotecan | Part 2: Irinotecan | Part 2: Topotecan
Number analyzed (Participants) | 187 | 190 | 94
months | 3.5 [2.8 to 4.2] | 3.0 [2.7 to 4.2] | 3.4 [2.8 to 4.2]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR is the percentage of subjects with best overall response of either complete response (CR) or partial response (PR); ORR = CR + PR. Per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, CR was defined as the disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters as confirmed by CT or MRI.
Time Frame: Up to approximately 2.5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Dinutuximab + Irinotecan | Part 2: Irinotecan | Part 2: Topotecan
Number analyzed (Participants) | 187 | 190 | 94
Participants | 32 | 36 | 19

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The CBR is defined as the percentage of subjects with either a CR, PR, or stable disease (SD), relative to the number of subjects in the treatment group. Per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, CR was defined as the disappearance of all target lesions; PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters; and SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study, as confirmed by CT or MRI .
Time Frame: Up to approximately 2.5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Dinutuximab + Irinotecan | Part 2: Irinotecan | Part 2: Topotecan
Number analyzed (Participants) | 187 | 190 | 94
Participants | 126 | 112 | 64

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for all enrolled subjects beginning with first dose of study medication. Serious adverse events (and AEs based on local regulations) were to be collected starting on the day of written informed consent. In addition to reporting while on study therapy, adverse events were required to be reported through 30 days after the last dose of study therapy.
Description: AEs were collected via Investigator assessment and laboratory testing during routine visits as required per protocol.
  For the analyses, All-Cause Mortality was evaluated for all subjects enrolled in Part 1 or randomized in Part 2 of the study and assigned treatment (n = 483). All other Safety Analyses, including Serious Adverse Events and Other Adverse Events, were evaluated using the Safety Analysis Set, defined as all subjects who received at least 1 dose of study medication (n = 470).
Arm/Group | Part 1: Dinutuximab + Irinotecan | Part 2: Dinutuximab + Irinotecan | Part 2: Irinotecan | Part 2: Topotecan
All-Cause Mortality (participants affected / at risk) | 10/12 | 158/187 | 159/190 | 84/94
Serious Adverse Events (participants affected / at risk) | 5/12 | 74/183 | 76/187 | 39/88
Other Adverse Events (participants affected / at risk) | 12/12 | 183/183 | 183/187 | 86/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Dinutuximab + Irinotecan (N=12) | Part 2: Dinutuximab + Irinotecan (N=183) | Part 2: Irinotecan (N=187) | Part 2: Topotecan (N=88)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 8 | 17 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 7 | 7 | 4
Anemia (Blood and lymphatic system disorders) | 0 | 4 | 2 | 6
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 8 | 17 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 7
Bradycardia (Cardiac disorders) | 0 | 2 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Endocarditis noninfective (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 6 | 9 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 4 | 1 | 1
Chest pain (General disorders) | 0 | 2 | 0 | 0
Pain (General disorders) | 0 | 2 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0
General physical health deterioration (General disorders) | 0 | 0 | 5 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 6 | 9 | 5
Sepsis (Infections and infestations) | 0 | 3 | 3 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 2 | 0
Septic shock (Infections and infestations) | 1 | 1 | 3 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 4 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis pseudomonas (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 2 | 4 | 3
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 5
Troponin I increased (Investigations) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 5 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 2 | 1 | 0
Syncope (Nervous system disorders) | 0 | 2 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 1 | 0
Neurological decompensation (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 4
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 3 | 2 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
Superior vena cava occlusion (Vascular disorders) | 0 | 0 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Dinutuximab + Irinotecan (N=12) | Part 2: Dinutuximab + Irinotecan (N=183) | Part 2: Irinotecan (N=187) | Part 2: Topotecan (N=88)
Anaemia (Blood and lymphatic system disorders) | 3 | 67 | 55 | 58
Neutropenia (Blood and lymphatic system disorders) | 4 | 59 | 47 | 45
Leukopenia (Blood and lymphatic system disorders) | 0 | 30 | 22 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 18 | 13 | 22
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 11 | 18 | 4
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 118 | 116 | 13
Abdominal pain (Gastrointestinal disorders) | 5 | 82 | 24 | 9
Nausea (Gastrointestinal disorders) | 7 | 81 | 88 | 22
Vomiting (Gastrointestinal disorders) | 5 | 65 | 57 | 6
Abdominal pain upper (Gastrointestinal disorders) | 2 | 30 | 11 | 5
Constipation (Gastrointestinal disorders) | 4 | 16 | 16 | 13
Dysphagia (Gastrointestinal disorders) | 1 | 6 | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 4 | 4 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 4 | 9 | 6
Abdominal pain lower (Gastrointestinal disorders) | 1 | 3 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 3 | 4 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Asthenia (General disorders) | 4 | 44 | 39 | 25
Fatigue (General disorders) | 3 | 36 | 48 | 16
Non-cardiac chest pain (General disorders) | 1 | 24 | 8 | 5
Pyrexia (General disorders) | 2 | 19 | 10 | 13
Pain (General disorders) | 0 | 13 | 5 | 1
Chest pain (General disorders) | 1 | 11 | 5 | 1
Chest discomfort (General disorders) | 1 | 5 | 2 | 0
Discomfort (General disorders) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 12 | 11 | 9
Upper respiratory tract infection (Infections and infestations) | 1 | 5 | 10 | 2
Septic shock (Infections and infestations) | 1 | 2 | 3 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 3 | 3
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 4 | 0
Weight decreased (Investigations) | 1 | 24 | 25 | 8
Blood lactate dehydrogenase increased (Investigations) | 0 | 19 | 6 | 5
Neutrophil count decreased (Investigations) | 1 | 18 | 28 | 23
Alanine aminotransferase increased (Investigations) | 0 | 12 | 13 | 8
Aspartate aminotransferase increased (Investigations) | 0 | 10 | 11 | 8
Platelet count decreased (Investigations) | 1 | 10 | 6 | 18
Blood alkaline phosphatase increased (Investigations) | 0 | 7 | 6 | 5
White blood cell count decreased (Investigations) | 0 | 6 | 12 | 14
Lymphocyte count decreased (Investigations) | 0 | 5 | 4 | 5
Blood creatinine increased (Investigations) | 1 | 3 | 4 | 1
Clostridium test positive (Investigations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 5 | 60 | 58 | 23
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 18 | 16 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 14 | 17 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 10 | 14 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 8 | 4 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 7 | 9 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 6 | 11 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 6 | 3 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 47 | 11 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 31 | 5 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 16 | 8 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 13 | 3 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 12 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 11 | 2 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 10 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 2
Headache (Nervous system disorders) | 2 | 21 | 12 | 4
Dizziness (Nervous system disorders) | 0 | 12 | 15 | 6
Neuropathy peripheral (Nervous system disorders) | 2 | 3 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 6 | 2 | 2
Confusional state (Psychiatric disorders) | 1 | 3 | 2 | 2
Agitation (Psychiatric disorders) | 1 | 0 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 28 | 16 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 27 | 18 | 13
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 11 | 6 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 8 | 4 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 49 | 33 | 10
Rash (Skin and subcutaneous tissue disorders) | 2 | 4 | 4 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 15 | 9 | 5
Hypertension (Vascular disorders) | 1 | 14 | 4 | 3
Flushing (Vascular disorders) | 1 | 4 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submission for any public disclosure of the data or results, the Institution and Principal Investigator shall provide Sponsor with at least 60 days for review of the Publication. In addition, the Institution and Principal Investigator agree that the first Publication of the results shall be made as a joint, multicenter publication coordinated by Sponsor, with investigators and institutions from all participating sites contributing data.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-12-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT03098030/SAP_000.pdf
  • Study Protocol (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT03098030/Prot_001.pdf